CLINICAL TRIAL: NCT01636193
Title: Drug Use Investigation for ROTARIX
Brief Title: Drug Use Investigation for ROTARIX®
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115926
Record Dates: First submitted 2012-06-25; First posted 2012-07-10 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus; Rotarix; Drug Use Investigation; Safety
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rota Group: Subjects will receive Rotarix® as per routine practice.
  Interventions: Biological: Oral Rotarix®; Other: Data collection

INTERVENTIONS:
Biological: Oral Rotarix® — 2 doses administered orally.
Other: Data collection — Safety data will be collected through the check of health observation diary and interview of vaccinee's parent.

SUMMARY:
This study aims to assess the safety of Oral Rotarix® under clinical practice; and collect information regarding typical symptoms of intussusceptions and bloody stool in Japan.

DETAILED DESCRIPTION:
This is non-interventional study conducted in one group received Oral Rotarix®. This surveillance is abbreviated as SMILER (Surveillance and Monitoring In Living clinical Experience for Rotarix).

ELIGIBILITY:
Inclusion Criteria:

• Infants who receive Rotarix for the first time to prevent rotavirus gastroenteritis, an indication of Rotarix, will be included in the investigation.

Exclusion Criteria:

• All infants included in the special drug use investigation of Oral Rotarix will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants who receive Rotarix for the first time to prevent rotavirus gastroenteritis as part of routine immunisation programme.
Sampling Method: Non-Probability Sample
Enrollment: 1607 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse events under clinical practice. | During the 31-day observation period after each vaccination.
Occurrence of typical symptoms of intussusceptions and bloody stool. | During the 31-day observation period after each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline